CLINICAL TRIAL: NCT00610558
Title: Neocortical Epilepsies - Do They Progress?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Min-Ying (Lydia) Su, Professor, University of California, Irvine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UCI-HS-2003-3252; VA-821/103 (Other: VAMC West Los Angeles)
Record Dates: First submitted 2008-01-12; First posted 2008-02-08 (Estimated); Results first posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: Three different Groups in this study: Juvenile Myoclonic Epilepsy, Frontal Lobe Epilepsy, Normal Controls
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1: Juvenile Myoclonic Epilepsy (Experimental): Juvenile Myoclonic Epilepsy group of subjects will participate for imaging assessment
  Interventions: Device: Arm 1: Juvenile Myoclonic Epilepsy
- Arm 2: Frontal Lobe Epilepsy (Experimental): Frontal Lobe Epilepsy group of subjects will participate for imaging assessment
  Interventions: Device: Arm 2: Frontal Lobe Epilepsy
- Arm 3: Normal Controls (Experimental): Normal Controls, eligible subjects don't have Juvenile Myoclonic Epilepsy or Frontal Lobe Epilepsy will be placed in this group
  Interventions: Device: Arm 3: Normal Controls

INTERVENTIONS:
Device: Arm 1: Juvenile Myoclonic Epilepsy — Positron emission tomography (PET) fluorodeoxyglucose (FDG) (10 mCi) and MRI
  Arms: Arm 1: Juvenile Myoclonic Epilepsy
Device: Arm 2: Frontal Lobe Epilepsy — Positron emission tomography (PET) fluorodeoxyglucose (FDG) (10 mCi) and MRI
  Arms: Arm 2: Frontal Lobe Epilepsy
Device: Arm 3: Normal Controls — Positron emission tomography (PET) fluorodeoxyglucose (FDG) (10 mCi) and MRI
  Arms: Arm 3: Normal Controls

SUMMARY:
This study will use MRI and PET scan to compare the brain imaging results between epilepsy patients and normal healthy controls, also to study changes in 3 years.

DETAILED DESCRIPTION:
We would like to continue analyzing the structural and metabolic differences between two epilepsy groups (JME and FLE) and the control to understand the imaging presentations of epilepsy patients

ELIGIBILITY:
Controls (20 Subjects):

Inclusion criteria:

* Ages 18-65, based on the usual ages of patients seen in the adult neurology services who are not likely to suffer from the exclusions (see below).

Exclusion criteria:

* History of seizures, faints, or any unexplained blackouts.
* Use of neuroleptic medications or sedating doses of antianxiety or antidepressant drugs.
* They should not have a clear family history of epilepsy (first degree relatives).
* History of any substance abuse within the past 5 years.
* History of progressive medical or neurologic disease (Parkinson's, severe congestive heart failure). Controlled hypertension, diabetes (by oral medications or diet), asthma, etc will not be excluded.
* History of stroke without complete recovery of neurologic function.
* Pregnancy
* With any metallic implants, including surgical clips (hemostatic clips), pacemakers, neuro-stimulation devices, prosthetic heart valves, or other ferromagnetic material.
* Inability to understand the consent. (standard form attached)
* Inability to speak fluent English. Note: the neuropsychological tests are standardized for English speakers. They are not all available in multiple languages. Since the scoring and norms are established for English speakers, simply translating them would still not make the testing norms and scoring applicable.

Juvenile Myoclonic Epilepsy (JME; 20 Subjects):

Inclusion Criteria:

* Ages 18-65, based on the usual ages of patients seen in the adult neurology services who are not likely to suffer from the exclusions (see below), plus
* History of myoclonic plus tonic-clonic or clonic-tonic-clonic seizures with or without absence seizures.
* EEG consistent with primary generalized epilepsy (>/= 3 c/s generalized, frontal maximum, poly spike and wave; normal alpha)

Exclusion Criteria

* History of significant head injury (> 30 min loss of consciousness)
* Use of neuroleptic drugs or sedative doses of antianxiety or antidepressant drugs
* History of any substance abuse within the past 5 years
* Presence of epileptogenic brain lesion on MRI (tumor, stroke, cortical congenital dysplasia, etc; excluding normal variants, mild subcortical white matter ischemic change, venous angiomas).
* EEG with focal epileptiform potentials or polymorphic slowing
* History of progressive medical or neurologic disease (Parkinson's, severe congestive heart failure). Controlled hypertension, diabetes (by oral medications or diet), asthma, etc will not be excluded.
* History of stroke without complete recovery of neurologic function.
* Pregnancy
* With any metallic implants, including surgical clips (hemostatic clips), pacemakers, neuro-stimulation devices, prosthetic heart valves, or other ferromagnetic material.
* Inability to speak fluent English

Frontal Lobe Epilepsy (FLE; 20 Subjects):

Inclusion Criteria

* Ages 18-65, based on the usual ages of patients seen in the adult neurology services who are not likely to suffer from the exclusions (see below), plus:
* Seizure semiology (behavior) consistent with FLE
* Interictal EEG spikes consistent with FLE or
* Ictal video-EEG consistent with FLE
* Frontal lobe lesion of MRI
* Frontal hypometabolism on FDG-PET

Exclusion Criteria:

* Presence of seizure semiology, ictal EEG, interictal EEG, MRI or PET findings that are not consistent with a frontal lobe epilepsy focus.
* Use of neuroleptic drugs or sedative doses of antianxiety or antidepressant drugs
* History of any substance abuse within the past 5 years
* History of progressive medical or neurologic disease (Parkinson's, severe congestive heart failure). Controlled hypertension, diabetes (by oral medications or diet), asthma, etc will not be excluded.
* History of stroke without complete recovery of neurologic function.
* Pregnancy
* With any metallic implants, including surgical clips (hemostatic clips), pacemakers, neuro-stimulation devices, prosthetic heart valves, or other ferromagnetic material.
* Absence of either a radial or ulnar arterial pulse
* Inability to speak fluent English

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2003-07; Primary Completion 2009-06 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Min-Ying Su, PhD, Principal Investigator — University of California, Irvine
Locations (1):
- Center for Functional Onco-Imaging, University of California, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There is no pre-assignment for this study
Groups:
- Arm 1: Juvenile Myoclonic Epilepsy; Arm 2: Frontal Lobe Epilepsy; Arm 3: Normal Cont: Subjects who are eligible for this group will participate MRI imaging
Period: Overall Study
Arm/Group | Arm 1: Juvenile Myoclonic Epilepsy | Arm 2: Frontal Lobe Epilepsy | Arm 3: Normal Cont
Started | 20 | 20 | 20
Completed | 15 | 14 | 14
Not Completed | 5 | 6 | 6

BASELINE CHARACTERISTICS:
Population: The imaging data of Arm 3 will be the baseline to compare the difference to the imaging data in Arm 1 and Arm 2. We used an MRI-based with high angular resolution imaging examination of adult human brains. We compared the connectivity patterns in control subjects versus patients with Juvenile Myoclonic Epilepsy or Frontal Lobe Epilepsy,
Groups:
- Arm1: Juvenile Myoclonic Epilepsy; Arm 2: Frontal Lobe Epilepsy; Arm 3: Normal Controls: Subject will are eligible for this group will participate the MRI imaging
- Total: Total of all reporting groups
Arm/Group | Arm1: Juvenile Myoclonic Epilepsy | Arm 2: Frontal Lobe Epilepsy | Arm 3: Normal Controls | Total
Number analyzed (Participants) | 15 | 14 | 14 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 14 | 14 | 43
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (6.5) | 37 (6.8) | 40 (7.7) | 38.3 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 7 | 23
  Male | 7 | 6 | 7 | 20
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 14 | 14 | 43

OUTCOME MEASURES:

1. Primary Outcome: Functional Connectivity
Description: We will analyze the structural and metabolic differences between two epilepsy groups (JME and FLE) and understand the imaging presentations of epilepsy patients. We will process imaging requisition for Arm 1 and Arm 2 patients and the controls to examine if any differences in their brain image. The hypothesis is the functional connectivity between brainstem structures and cortical/subcortical regions may reflect in their imaging data. We would like to know if these imaging factors are related to epilepsy (JME and FLE) patients.
Time Frame: During Imaging Session
Population: This protocol has been closed about 10 years ago. All files have been destroyed per IRB requirement.
Groups:
- Arm 1: Juvenile Myoclonic Epilepsy: Subjects who are eligible to Juvenile Myoclonic Epilepsy will participate the imaging study
- Arm 2: Frontal Lobe Epilepsy: Subjects who are eligible to Frontal Lobe Epilepsy will participate the imaging study
- Arm 3: Normal Controls: Subjects who are eligible to the control group will participate the imaging study
Arm/Group | Arm 1: Juvenile Myoclonic Epilepsy | Arm 2: Frontal Lobe Epilepsy | Arm 3: Normal Controls
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Subjects monitored for safety events during the entire imaging session; up to 1 hour
Description: All-Cause Mortality, Serious, and non-serious Adverse Events were monitored/assessed, but none observed
Groups:
- Arm 1: Juvenile Myoclonic Epilepsy: 15 Subjects were monitored/assessed, but none observed
- Arm 2: Frontal Lobe Epilepsy; Arm 3: Normal Controls: 14 Subjects were monitored/assessed, but none observed
Arm/Group | Arm 1: Juvenile Myoclonic Epilepsy | Arm 2: Frontal Lobe Epilepsy | Arm 3: Normal Controls
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/15 | 0/14 | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Juvenile Myoclonic Epilepsy (N=15) | Arm 2: Frontal Lobe Epilepsy (N=14) | Arm 3: Normal Controls (N=14)
Allergic reactions to the contrasts (General disorders) | 0 (0) | 0 (0) | 0 (0) — Allergic reactions to the radiopharmaceutical may occur, but are extremely rare.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Juvenile Myoclonic Epilepsy (N=15) | Arm 2: Frontal Lobe Epilepsy (N=14) | Arm 3: Normal Controls (N=14)
Bleeding, soreness or swelling of injection site (General disorders) | 0 (0) | 0 (0) | 0 (0) — Bleeding, soreness or swelling may develop at injection site.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No